CLINICAL TRIAL: NCT06597318
Title: Trends of Patient-reported Outcome Measures (PROMs) in Multimorbid Medical Patients Hospitalized for an Acute Illness
Acronym: TRADUCE
Status: Recruiting | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); University Hospital, Zürich (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Marie Méan, Principal Investigator, Senior Physician, University of Lausanne Hospitals
Other Study IDs: 2023-00200
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PROM; PREM; Quality of Care; Internal Medicine
MeSH Terms: interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multimorbid patients in general internal medicine divisions of all five Swiss university hospitals
  Interventions: Other: Hospitalization

INTERVENTIONS:
Other: Hospitalization — The investigators collect PROMs amongst up to 1000 patients in general internal medicine divisions of all five Swiss university hospitals

SUMMARY:
currently, PROMs and PREMs are not routinely collected and compared among medical inpatients of Swiss university hospitals, nor is a standard set of PROMs and PREMs available for use in Swiss hospitals. The project aims to examine trends in patient-reported outcomes (PROMs), including symptoms, quality of life, and distress, in multimorbid hospitalized patients from admission to 30 days post-discharge. It will also investigate whether PROMs at discharge are linked to the risk of readmission or emergency visits and explore how these outcomes differ in patients who receive low-value care. Additionally, the project will assess the relationship between patient-reported experiences (PREMs) and the provision of low-value care during the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* eligible for the LUCID registry (CER-VD AO_2023-00029) [Age ≥ 18 years, hospitalized in one of the five participating university hospitals (Geneva, Lausanne, Bern, Zürich, Basel), after 01.01.2014, and admitted to general internal medicine wards
* Multimorbid patients (2 or more chronic diseases, defined as chronic conditions defined by international classification of diseases, 10th revision, codes with an estimated expected duration of at least 6 months or based on a clinical decision.
* Acute illness
* Signature of study specific informed consent

Exclusion Criteria:

* Not able to speak French, German or English
* Foreseen length of stay of less than 4 days (estimated by study collaborators)
* Prior inclusion in the TRADUCE study
* Incapacity of discernment, i.e. cognitive impairment which could interfere with the ability to fill in PROMs tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 2 or more chronic diseases, hospitalized in general internal medicine divisions of all five Swiss university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of PROMS with the risk of readmission | Day 1, Day 3, at the day of discharge (approximately day 8) and Day 30 after discharge from Hospital
  The primary objective of the project is to explore trends in PROMs (using the Edmonton Symptom Assessment System (ESAS-r), the EQ-5D-5L index,45 and the National Comprehensive Cancer Network (NCCN) distress thermometer) of multimorbid medical hospitalized patients, from admission until 30-days post-discharge. The patients-reported outcomes will consist of patients-reported symptoms, quality of life and distress

SECONDARY OUTCOMES:
Correlation of PROMs at discharge and risk of hospital readmission or ED visits | Day 30 after discharge from hospital
  assess whether PROMs ((using the Edmonton Symptom Assessment System (ESAS-r), the EQ-5D-5L index,45 and the National Comprehensive Cancer Network (NCCN) distress thermometer) at discharge are associated with the risk of hospital readmission or of emergency department visit within the next 30 days;
Exploration of PROMs in patients who receive low-value care | Day 1, Day 3, at the day of discharge (approximately day 8) and Day 30 after discharge from Hospital
  explore whether PROMs ((using the Edmonton Symptom Assessment System (ESAS-r), the EQ-5D-5L index,45 and the National Comprehensive Cancer Network (NCCN) distress thermometer) trends vary in patients who do or do not receive low value care (LVC);
Explore PREMs | Since 24 hours after beginning of the hospitalization up to Discharge from Hospital (approximately day 8)
  Explore information on Patient Reported Experiences Measures (PREMs) using a qualitative questionnaire during patients' stay at the hospital, and whether there is a correlation between the provision of LVC and qualitative analysis of PREMs

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Stirnemann, MD, Principal Investigator — University Hospital, Geneva; Carole Aubert, MD, Principal Investigator — Bern University Hospital; Florence Vallelian Cervetto, MD, Principal Investigator — Zürich University Hospital; Stefano Bassetti, MD, Principal Investigator — Basel University Hospital
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No